CLINICAL TRIAL: NCT06713460
Title: Assessment of a Multicomponent Intervention Based on Emotional Intelligence to Improve Mental Well-being in Adolescents With Emotional Distress: A Randomized Controlled Trial
Brief Title: Emotional Intelligence Intervention to Improve Mental Well-Being of Adolescents With Emotional Distress (BEAM)
Acronym: BEAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, Maria Llistosella, Principal Investigator, Consorci Sanitari de Terrassa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 01-24-1CR-102
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Emotional Distress
Keywords: Mental Well-being; Emotional Intelligence; Emotional Distress; Adolescents
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the control or intervention group by an external investigator through computer-generated random numbers.
Masking Description: Due to the difficulty of masking conditions, the groups and participating personnel (research team) will not be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (multicomponent intervention) (Experimental): A multi-component group intervention, based on Mayer and Salovey's emotional skills model, will target adolescents with emotional distress. Led by the Community Emotional Well-Being Coordinator and supported by a nurse, physiotherapist, and educational psychologist, the intervention will occur April and November 2025 in Consorci Sanitari de Terrassa institutes. It will consist of nine 55-minute sessions during school hours, supplemented by voluntary home activities. The program will focus on emotional identification and regulation, structured around seven components: goal-setting, positive thinking, self-awareness, self-esteem, willpower, mindfulness, and assertiveness.
  Interventions: Behavioral: BEAM
- Control group (non intervention) (No Intervention): Participants in the control group will complete the same research questionnaires as the intervention group during the same period April and November 2025 Control group participants will undergo the intervention (if effective) in the following academic year (January - June 2026), when they are in 10th Grade.

INTERVENTIONS:
Behavioral: BEAM — Multicomponent intervention
  Arms: Intervention group (multicomponent intervention)

SUMMARY:
The goal of this clinical trial is to assess the effectiveness of a multicomponent intervention in adolescents with emotional distress. The main question it aims to answer is:

Does the intervention increase mental well-being, emotional resilience, and emocional intelligence in adolescents with emotional distress?

Participants will:

• Participate in a multi-component intervention for 9 weeks at school.

DETAILED DESCRIPTION:
Background:Adolescence involves biological, psychological and social transformations that increase vulnerability to mental health problems. Emotional intelligence is a protective factor that improves mental well-being. Given the sensitivity of adolescence to mental health disorders, emotional intelligence emerges as a valuable tool for promoting mental well-being.The investigators hypothesize that adolescents aged 14-16 with emotional distress who receive the multicomponent intervention based on emotional intelligence will obtain better scores on the Warwick-Edinburgh Mental Well-being Scale compared to the control group, after the intervention and at 24 weeks post-intervention.

Method :The study is a Randomized Controlled Trial (RCT). The participants and their parents will sign an agreement to participate in the study and will be randomly allocated in control and intervention groups by external researcher using a computer-generated random number. The intervention will be conducted in a school setting between April and November 2025. It will comprise a multicomponent program consisting of nine sessions, each lasting 55 minutes, addressing various topics related to emotional intelligence. Data will be collected from April 2025 to April 2026."Three psychometric scales will be used: Warwick-Edinburgh Mental Wellbeing Scale (WEMWB), Trait Meta-Mood Scale (TMMS-24) and Child Youth Resilience Measure (CYRM-32), with measurements before the intervention (T0), 9 (T1) and 24 weeks follow-up (T2).The group receiving the intervention is expected to show improvements in emotional well-being, emotional intelligence and resilience compared to the control group.

Accepting an alpha risk of 0.05 and a beta risk of 0.20 in a bilateral contrast, 52 subjects in the first group and 52 in the second group are required to detect a difference equal to or greater than 5 units on the WEMWBS scale. A common standard deviation of 6.8 is assumed. A loss to follow-up rate of 0.1 (10%) and a correlation between observations of 0.4 was estimated.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents with emotional distress scores on the Warwick-Edinburgh Mental Well- being Scale.
* Adolescents aged 14-16 ( in 9th Grade).
* Informed consent form signed (by adolescents and their parent or legal guardian)

Exclusion Criteria:

* Physical illnesses that prevent attendance at scheduled sessions, severe mental disorders (such as Autism Spectrum Disorder, major depression, schizophrenia).
* No comprehension of the language
* Lack of consent from the adolescents or their parents or legal guardians

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 104 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Improve well-being | Baseline (T0), post-intervention (9 weeks) (T1), and 24 weeks follow-up (T2)
  Changes in level of well-being using the Warwick-Edinburgh Mental Well-Being Scale (WEMWBS). Values range from 14 to 70 . Higher scores, better outcome.

SECONDARY OUTCOMES:
Increased resilience | Baseline (T0), post-intervention (9 weeks) (T1), and 24 weeks follow-up (T2)
  Changes in level of resilience using the Child Youth Resilience Measure -32. Values range from 32 to 160 . Higher scores, better outcome.
Increase emotional intelligence | Baseline (T0), post-intervention (9 weeks) (T1), and 24 weeks follow-up (T2)
  Changes in level of emotional intelligence using the Trait Meta-Mood Scale (TMMS). The TMMS-24 contains three key dimensions of EI with 8 items each: Emotional Attention: Adequate values: Males (22 to 32); Females (25 to 35); Emotional clarity: excellent values: Males (> 36); Females (>35), and Emotional repair: excellent values: Men (> 36); Women (>35)).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Llistosella, PhD, Principal Investigator — Primary Health Care, Consorci Sanitari de Terrassa
Locations (2):
- Spain (2):
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Institut Can Roca, Terrassa, Barcelona

IPD SHARING:
Plan to Share IPD: No
Fully anonymised overall results will be shared.

REFERENCES:
- [Background] Gracia R, Pamias M, Mortier P, Alonso J, Perez V, Palao D. Is the COVID-19 pandemic a risk factor for suicide attempts in adolescent girls? J Affect Disord. 2021 Sep 1;292:139-141. doi: 10.1016/j.jad.2021.05.044. Epub 2021 May 27. PMID 34119869
- [Result] Llistosella M, Gutierrez-Rosado T, Rodriguez-Rey R, Liebenberg L, Bejarano A, Gomez-Benito J, Limonero JT. Adaptation and Psychometric Properties of the Spanish Version of Child and Youth Resilience Measure (CYRM-32). Front Psychol. 2019 Jun 28;10:1410. doi: 10.3389/fpsyg.2019.01410. eCollection 2019. PMID 31316419
- [Result] Salguero, J. M., Fernández-Berrocal, P., Balluerka, N., & Aritzeta, A. (2010). Measuring perceived emotional intelligence in the adolescent population: Psychometric properties of the Trait Meta-Mood Scale. Social Behavior and Personality: an international journal, 38(9), 1197-1209
- [Result] Castellvi P, Forero CG, Codony M, Vilagut G, Brugulat P, Medina A, Gabilondo A, Mompart A, Colom J, Tresserras R, Ferrer M, Stewart-Brown S, Alonso J. The Spanish version of the Warwick-Edinburgh mental well-being scale (WEMWBS) is valid for use in the general population. Qual Life Res. 2014 Apr;23(3):857-68. doi: 10.1007/s11136-013-0513-7. Epub 2013 Sep 5. PMID 24005886
- [Result] Dominguez-Garcia E, Fernandez-Berrocal P. The Association Between Emotional Intelligence and Suicidal Behavior: A Systematic Review. Front Psychol. 2018 Nov 30;9:2380. doi: 10.3389/fpsyg.2018.02380. eCollection 2018. PMID 30555393